CLINICAL TRIAL: NCT00926042
Title: TAP0307: Enrollment of Normal Control Subjects for Current and Future Research
Brief Title: Genotype and Phenotype Registry: Enrollment of Normal Control Subjects for Current and Future Research
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Peter Gregersen, Center Head, Northwell Health
Other Study IDs: 04-007
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Healthy; volunteer; Healthy controls; Normal controls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek cell DNA sample will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Control: Healthy control group for research on autoimmune diseases

SUMMARY:
Registry program for volunteers who are willing to serve as control subjects in future research studies.

DETAILED DESCRIPTION:
The registry is a collection of volunteers willing to participate as control subjects in research studies. Control subjects are people who do not have a specific disease; therefore they can serve a critical role as a comparison with people who have the disease or other characteristic being studied. Once registered, participants will be notified about studies they may be able to participate in as a control.

Participation requires:

1. signing a consent form
2. answering a short health survey
3. providing a DNA sample via a mouthwash kit

The registry allows scientists to select study participants based on whether or not they have a specific genetic change that may be relevant to a disease under investigation. Having the ability to access controls when needed is an extremely valuable resource that will speed up scientific discoveries.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* over age 18

Exclusion Criteria:

* under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York City/ Long Island metropolitan community
Sampling Method: Non-Probability Sample
Enrollment: 4511 (Actual)
Dates: Start 2004-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Gregersen, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
available upon application and approval